CLINICAL TRIAL: NCT02184754
Title: Magnetic Endoscope Imaging in Single-balloon-enteroscopy
Acronym: Magenta
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 12-2014
Record Dates: First submitted 2014-01-02; First posted 2014-07-09 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Magnetic Endoscope Imaging in Single-balloon-enteroscopy
Keywords: Magnetic endoscope imaging; single-balloon-enteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MEI
  Interventions: Procedure: Magnetic endoscope imaging (MEI)

INTERVENTIONS:
Procedure: Magnetic endoscope imaging (MEI)
  Other Names: Olympus MAJ-Y0158

SUMMARY:
Magnetic endoscope imaging (MEI) is already used in colonoscopy in order facilitate scope navigation. In this study the use of MEI will be evaluated for small bowel enteroscopy in which scope navigation is particularly important. The MEI will be compared with x-ray which is still the current gold standard for scope navigation in small bowel enteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* indication for enteroscopy

Exclusion Criteria:

* contraindication for enteroscopy
* patients with cardiac pacemaker or defibrillator
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: endoscopy unit
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of concordance of MEI- and x-ray-images | 5 days
  Immediately after each examination MEI-images and x-ray-images will be analyzed for concordance

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, München, Bavaria, Germany